CLINICAL TRIAL: NCT05578573
Title: Comparison of Success Rate and Complication Between Conventional Angiocatheter Versus New Anchoring Device (KARAHOC) Used for Paracentesis in Cirrhotic Patients With Ascites
Brief Title: Comparison Between Conventional Angiocatheter Versus New Anchoring Device (KARAHOC) Used for Paracentesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sang Gyune Kim (Other)
Responsible Party: Sponsor-Investigator, Sang Gyune Kim, Professor, Soonchunhyang University Hospital
Organization: Soonchunhyang University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KARAHOC STUDY
Record Dates: First submitted 2022-01-16; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Ascites Hepatic
Keywords: paracentesis; cirrhosis; ascites
MeSH Terms: conditions — Fibrosis; Ascites

STUDY DESIGN:
Intervention Model Description: multi-center, prospective, interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KARAHOC group (Experimental): A group of patients in which paracentesis will be performed using a KARAHOC device.
  Interventions: Device: KARAHOC device
- conventional group (Active Comparator): A group of patients in which paracentesis will be performed using an angiocatheter.
  Interventions: Device: Angiocatheter

INTERVENTIONS:
Device: KARAHOC device — After leaving a mark on the part where the puncture is to be performed using a pen, sterilization dressing are performed, local anesthesia is performed aseptic then ascites paracentesis by KARAHOC device.
  Arms: KARAHOC group
Device: Angiocatheter — After leaving a mark on the part where the puncture is to be performed using a pen, sterilization dressing are performed, local anesthesia is performed aseptic then ascites paracentesis by angiocatheter
  Arms: conventional group

SUMMARY:
Comparison of success rate and complication between conventional angiocatheter versus new anchoring device (KARAHOC) used for paracentesis in cirrhotic patients with ascites.

DETAILED DESCRIPTION:
This study is a multi-center, prospective, interventional study, in which subjects who meet the selection criteria are registered at each institution during the study period from the date of research approval. Regardless of the order, paracentesis using KARAHOC and conventional angiocatheter will be performed once in all patients. The criteria for successful paracentesis is set as 3L or more of ascites drainage. During paracentesis, albumin will be infused in all patients. Heart rate and blood pressure will be measured before the procedure and right after the completion of drainage, and 30 minutes later. The incidence of complications will be compared between two methods. In addition, patient and operator satisfaction will be investigated using a visual analogue scale.

ELIGIBILITY:
Inclusion Criteria:

* Adult over the age of 19
* Patients with pathological or clinical diagnosis of liver cirrhosis
* Patients with Grade 2 or higher grade of ascites as a complication due to portal hypertension
* Patients requiring periodic paracentesis
* Patients consent to this study

Exclusion Criteria:(If at least one of the following conditions apply)

* Patients with ascites due to peritoneal metastasis due to malignant tumor
* Patients with high bleeding risk (PT INR>3, PLT<30,000/mm3) difficult to perform ascites puncture
* Patients with hepatic encephalopathy or hepatorenal syndrome(HRS)
* Patients with severe cardiovascular disease, lung disease, or DIC
* Patients refusing paracentesis
* Patients who can control ascites using diuretics
* Pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of success rate between conventional angiocatheter versus KARAHOC device used for paracentesis | through study completion, an average of 1 year
  The criterion for successful paracentesis is defined as drainage of 3L or more at an initial attempt.

SECONDARY OUTCOMES:
comparison of complication rate | through study completion, an average of 1 year
  the frequency of bleeding, hypotension, acute kidney injury, infection
operator satisfaction for each procedure | through study completion, an average of 1 year
  measure the amount of satisfaction using visual analogue scales distributed from 1 to 10, higher score means better outcome
patient satisfaction for each procedure | through study completion, an average of 1 year
  measure the amount of satisfaction using visual analogue scales distributed from 1 to 10, higher score means better outcome
Number of Participants with repeated paracentesis | through study completion, an average of 1 year
  Whether to do paracentesis again due to initial failure or catheter dislocation

CONTACTS AND LOCATIONS:
Overall Officials: Sang gyune Kim, PhD, Principal Investigator — Soonchunhyang University Hospital
Locations (1):
- Soon Chun Hyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Iwakiri Y. Pathophysiology of portal hypertension. Clin Liver Dis. 2014 May;18(2):281-91. doi: 10.1016/j.cld.2013.12.001. Epub 2014 Feb 25. PMID 24679494
- [Background] Moore KP, Aithal GP. Guidelines on the management of ascites in cirrhosis. Gut. 2006 Oct;55 Suppl 6(Suppl 6):vi1-12. doi: 10.1136/gut.2006.099580. No abstract available. PMID 16966752
- [Background] Gentilini P, Casini-Raggi V, Di Fiore G, Romanelli RG, Buzzelli G, Pinzani M, La Villa G, Laffi G. Albumin improves the response to diuretics in patients with cirrhosis and ascites: results of a randomized, controlled trial. J Hepatol. 1999 Apr;30(4):639-45. doi: 10.1016/s0168-8278(99)80194-9. PMID 10207805
- [Background] Gines P, Arroyo V, Quintero E, Planas R, Bory F, Cabrera J, Rimola A, Viver J, Camps J, Jimenez W, et al. Comparison of paracentesis and diuretics in the treatment of cirrhotics with tense ascites. Results of a randomized study. Gastroenterology. 1987 Aug;93(2):234-41. doi: 10.1016/0016-5085(87)91007-9. PMID 3297907
- [Background] Quintero E, Gines P, Arroyo V, Rimola A, Bory F, Planas R, Viver J, Cabrera J, Rodes J. Paracentesis versus diuretics in the treatment of cirrhotics with tense ascites. Lancet. 1985 Mar 16;1(8429):611-2. doi: 10.1016/s0140-6736(85)92147-6. PMID 2857949
- [Background] Salerno F, Badalamenti S, Incerti P, Tempini S, Restelli B, Bruno S, Bellati G, Roffi L. Repeated paracentesis and i.v. albumin infusion to treat 'tense' ascites in cirrhotic patients. A safe alternative therapy. J Hepatol. 1987 Aug;5(1):102-8. doi: 10.1016/s0168-8278(87)80067-3. PMID 3655306

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT05578573/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT05578573/ICF_001.pdf